CLINICAL TRIAL: NCT04222257
Title: Short-course Antibiotic Regimen Compared to Conventional Antibiotic Treatment for Gram-positive Cocci Infective Endocarditis: Randomized Clinical Trial
Brief Title: Short-course Antibiotic Treatment in Gram-positive Cocci Infective Endocarditis
Acronym: SATIE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to reach the estimated sample size
Sponsor: Carmen Olmos Blanco (Other)
Responsible Party: Sponsor-Investigator, Carmen Olmos Blanco, Principal investigator, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SATIE
Record Dates: First submitted 2019-12-19; First posted 2020-01-09 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Endocarditis, Bacterial
Keywords: Infective endocarditis; short-course; antibiotic therapy
MeSH Terms: conditions — Endocarditis, Bacterial; Endocarditis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short course (Experimental): Patients allocated to this group will receive a short course of antibiotic therapy for 2 weeks.
  Interventions: Drug: Antibiotics
- Standard course (Active Comparator): Those patients allocated to continue with standard parenteral treatment will maintain the same antibiotic treatment for 4 to 6 weeks.
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: Antibiotics — Patients allocated to this group will receive a short course of antibiotic therapy for 2 weeks.
  Arms: Short course
Drug: Antibiotics — Patients allocated to continue with standard parenteral treatment will maintain the same antibiotic treatment for 4 to 6 weeks.
  Arms: Standard course

SUMMARY:
Background: it is well known that most serious complications of infective endocarditis (IE) appear in the so-called "critical phase" of the disease, which are the first days after diagnosis. Subsequently, the vast majority of patients who overcome this acute phase has a favourable evolution, and usually stay in the hospital for a long time only to complete antibiotic therapy.

In stable patients with adequate response to antibiotic treatment, without signs of persistent infection or metastatic foci such as spondylodiscitis, it is likely that a shorter antibiotic regimen would be an efficient and safe alternative, as has already been confirmed in patients with IE on tricuspid valves caused by a microorganism considered virulent such as S. aureus. This attractive alternative would improve patients' quality of life, save costs, and decrease the risk of complications related to the adverse effects of prolonged antibiotic treatment.

Objectives: to compare the incidence of the composite endpoint of all-cause mortality, unplanned cardiac surgery, symptomatic embolisms and relapses within 6 months after the inclusion between patients with IE caused by gram-positive cocci receiving a short-course of 2 weeks of antibiotic therapy and those patients receiving conventional antibiotic therapy (4-6 weeks).

Methodology: multicenter, prospective, randomized, controlled open-label, phase IV clinical trial. Sample: patients with IE caused by gram-positive cocci, having received at least 10 days of conventional antibiotic treatment, and at least 7 days after surgery when indicated, without clinical, analytical, microbiological or echocardiographic signs of persistent infection. Estimated sample size: 298 patients. Intervention: Control group: standard antibiotic therapy, according to ESC guidelines recommendations, for 4 to 6 weeks. Experimental group: short-course antibiotic therapy for 2 weeks. The prevalence of previously known risk factors for adverse events will be compared between the two groups to confirm that randomization have worked properly. The incidence of the composite endpoint of all-cause mortality, unplanned cardiac surgery, symptomatic embolisms and relapses within 6 months after the inclusion in the study will be prospectively registered and compared.

ELIGIBILITY:
Inclusion Criteria:

* Definite IE, according to modified ESC 2015 criteria, caused by gram-positive cocci (staphylococci, streptococci and enterococci), including native, prosthetic valve IE and cardiac device-related IE.
* 18 years old or older.
* Patients treated for at least 10 days of appropriate parenteral antibiotic therapy overall (according to guidelines and microbiology sensitivity testing), and at least 7 days of parenteral antibiotic therapy after valve surgery when indicated.
* Absence of fever, microbiological or analytical findings suggesting persistent infection at randomization.
* Absence of locally uncontrolled infection signs (abscess, pseudoaneurysm, fistula, enlarging vegetation) at randomization, confirmed by recent transesophageal echocardiography (performed within 48 h of randomization).
* Women of childbearing potential who will agree to the use of effective contraceptive methods while on antibiotic treatment.

Exclusion Criteria:

* Patients who have received appropriate parenteral antibiotic therapy for infective endocarditis for more than 12 days.
* Patients not suitable to be discharged after 10 days of conventional treatment, due to clinical reasons (sequels of stroke that prevent discharge, progressive renal failure, hepatic failure).
* Patients receiving chemotherapy or immunosuppressive therapy.
* Pregnant or breastfeeding women.
* Need of prolonged antibiotic therapy due to spondylodiscitis or other septic complication.
* Absence of patient's ability or commitment to continue follow-up after being discharged from hospital.
* Inability to give informed consent to participation.
* Cognitive impairment or lack of language skills needed to complete the questionnaires.
* Patients who meet urgent cardiac surgery ESC criteria but are considered inoperable due to high surgical risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Composite endopoint | 6 months
  To compare the incidence of the composite endpoint that includes all-cause mortality, unplanned cardiac surgery, symptomatic embolisms and relapses within 6 months after the inclusion, between patients with IE caused by gram-positive cocci receiving a short course of 2 weeks of antibiotic therapy and those patients receiving conventional antibiotic therapy for 4-6 weeks.

SECONDARY OUTCOMES:
Perceived quality of life: SF-12 | 4 weeks
  Determination of quality of life (SF-12)
Functional performance | 4 weeks
  Determination of functional performance according to the short performance physical battery test (SPPB)
Clinical complications | 6 months
  Clinical complications related to hospital stay (nosocomial infections, intravascular catheter-related infections)
Total hospital length of stay | 6 months
  Total hospital length of stay in the next 6 months after the inclusion in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Institute. Hospital Clínico San Carlos, Madrid, Spain

REFERENCES:
- [Derived] Olmos C, Vilacosta I, Lopez J, Saez C, Anguita M, Garcia-Granja PE, Sarria C, Silva J, Alvarez-Alvarez B, Martinez-Monzonis MA, Castillo JC, Seijas J, Lopez-Picado A, Peral V, Maroto L, San Roman JA. Short-course antibiotic regimen compared to conventional antibiotic treatment for gram-positive cocci infective endocarditis: randomized clinical trial (SATIE). BMC Infect Dis. 2020 Jun 16;20(1):417. doi: 10.1186/s12879-020-05132-1. PMID 32546269